CLINICAL TRIAL: NCT07079033
Title: Can We Reliably Needle Hip Region Muscles Without Imaging? A Muscle-Specific Accuracy Study Using Ultrasound
Brief Title: Can We Reliably Needle Hip Muscles Blindly?
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erzurum Regional Training & Research Hospital (Other Government)
Responsible Party: Principal Investigator, nurmuhammet tas, dr., Erzurum Regional Training & Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: erzurum rtrh2
Record Dates: First submitted 2025-06-23; First posted 2025-07-22 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Hip Needling
Keywords: dry needling; trigger point; ultrasound guidance

STUDY DESIGN:
Intervention Model Description: Dry needling is performed using anatomical landmarks without ultrasound guidance. Needle placement is then confirmed via ultrasound imaging.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blind Dry Needling Lumbar Paraspinal Muscles (Experimental): Dry needling is performed using anatomical landmarks without ultrasound guidance. Needle placement is then confirmed via ultrasound imaging.
  Interventions: Procedure: Blinded Dry Needling

INTERVENTIONS:
Procedure: Blinded Dry Needling — Dry needling is performed using anatomical landmarks without ultrasound guidance. Needle placement is then confirmed via ultrasound imaging.

SUMMARY:
The aim of this study is to evaluate the accuracy of invasive interventions (dry needling or injection) performed on specific muscles of the hip region in reaching the anatomical target. The accuracy of the interventions performed with a blinded method will be compared with an observational assessment supported by ultrasonography. The interventions will be performed by a physician with clinical experience, and the anatomical location of the needle tip will be evaluated by a second physician with ultrasonography after each procedure. The targeted muscles include the iliacus, pectineus, sartorius, tensor fascia latae, and rectus femoris. Each participant will be subjected to interventions for five different muscles, and a total of at least 40 injection interventions will be analyzed. Ultrasonography will be used only for observation and verification purposes; no pharmacological substances will be applied during the procedure. All procedures will be performed under sterile conditions, and participants will be monitored for 24 hours for possible pain, bruising, or complications. Participants will be informed about the content and purpose of the study, and written informed consent forms will be obtained. The study does not have a therapeutic purpose and is only intended to investigate targeting accuracy. The data to be obtained is expected to contribute to the determination of anatomical accuracy rates in clinical practices and the improvement of interventional training processes.

DETAILED DESCRIPTION:
This study aims to evaluate the accuracy of muscle targeting when dry needling injections are performed using the blinded (anatomical landmark-based) technique. The accuracy of these injections will be assessed by confirming the needle placement with ultrasonography immediately after each attempt.

According to existing literature, the accuracy of blinded injection techniques is reported to be approximately 67%, while ultrasound-guided injections achieve an accuracy of about 92%. A power analysis was conducted using these proportions to detect a statistically significant difference between the two methods. Based on these values, Cohen's h effect size was calculated as 0.66. With a significance level (alpha) of 0.05 and a statistical power of 80%, a minimum of 74 injection attempts are required.

In this study, each participant will receive injections into five different muscles suspected to be involved in myofascial pain. With 15 participants, this will result in 75 injection attempts, thereby meeting the required sample size for adequate power.

Eligible participants will be adults aged 18-65 presenting with nonspecific hip, groin, or anterior thigh pain and referred for physical therapy. The study particularly focuses on individuals with suspected myofascial pain syndrome in deep or less accessible hip-related muscles, such as the iliacus, pectineus, and sartorius. All participants must be clinically indicated for dry needling or similar interventions and capable of cooperating with the procedure.

Ultrasonographic evaluation will be used only to confirm needle placement, not to guide the injection. This allows for the assessment of the real-world accuracy of the blinded technique, which is commonly used in routine clinical practice. The findings will provide insight into the reliability of this method and help guide training and clinical decision-making in musculoskeletal and pain management practices.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65 years
* Individuals with nonspecific hip, groin, or anterior thigh pain who are scheduled for physical therapy
* Clinical suspicion of myofascial pain syndrome, particularly involving muscles around the hip
* Patients with clinical indication for dry needling or similar invasive treatments (e.g., targeting muscles such as iliacus, pectineus, sartorius)
* Ability to cooperate with the procedure
* Ability to provide written informed consent

Exclusion Criteria:

* Use of anticoagulant medications (due to increased risk of bleeding)
* Severe hip osteoarthritis, presence of hip prosthesis, history of previous hip surgery, or significant anatomical deformity
* Active infection or skin lesion at the planned injection site
* Inability to cooperate or communicate effectively
* Pregnancy
* Presence of serious systemic illnesses (e.g., malignancy, neurological disorders)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-28 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Blinded Dry Needling Injections | Immediately after each injection attempt
  Proportion of injection attempts in which the needle accurately reaches the intended target muscle using the blinded (anatomical landmark-based) technique, as confirmed by ultrasonography.

SECONDARY OUTCOMES:
Accuracy Rate per Target Muscle | Immediately after each injection attempt
  Determination of individual accuracy rates for each of the five specific muscles injected using the blinded technique (e.g., iliacus, pectineus, sartorius, etc.), based on ultrasound confirmation.

OTHER OUTCOMES:
Inter-Operator Variability in Injection Accuracy | 2 week
  Evaluation of variability in injection accuracy among different clinicians performing the blinded technique, based on ultrasound-confirmed needle placements.

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD) from this study.